CLINICAL TRIAL: NCT04568681
Title: Deep Brain Stimulation Effects in Dystonia: Time Course of Electrophysiological Changes in Treatment
Brief Title: Deep Brain Stimulation Effects in Dystonia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202002270
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with dystonia: Patients with dystonia who have clinically been deemed candidates for DBS surgery.
  Interventions: Device: Deep brain stimulation (DBS)

INTERVENTIONS:
Device: Deep brain stimulation (DBS) — Deep brain stimulation is an FDA approved therapy that involves surgical implantation of electrodes in deep brain targets and an implantable pulse generator delivers electrical pulses.

SUMMARY:
Deep Brain Stimulation (DBS) is an effective therapy for patients with medically refractory primary dystonia. However, DBS programming for dystonia is not standardized and multiple clinic visits are frequently required to adequately control symptoms. We aim to longitudinally record brain signals from patients using a novel neurostimulator that can record brain signals. We will correlate brain signals to clinical severity scores to identify pathological rhythms in the absence of DBS, and we will study the effects of DBS on these signals in order to guide clinical programming. We are going to recruit patients who receive the Medtronic Percept device, which allows for brain signal recordings (this feature is FDA approved). The investigators will be conducting an observational study using this device to collect data that the subjects receive as standard of care.

DETAILED DESCRIPTION:
The development of newer technologies has allowed clinicians and researchers to better understand pathophysiological underpinnings of different disorders managed with neuromodulation. There is a paucity of information, however, on dystonia, likely due to its rarity of cases and variability in phenomenology to allow generalization of findings. Possible abnormal brain signals, such as high activity in theta band (defined as rhythms in the 4-12Hz range ), have been proposed by small case series. The development of newer technologies has allowed clinicians and researchers to better understand pathophysiological underpinnings of different disorders managed with neuromodulation. There is a paucity of information, however, on dystonia, likely due to its rarity of cases and variability in phenomenology to allow generalization of findings. Possible abnormal brain signals, such as high activity in theta band (defined as rhythms in the 4-12Hz range ), have been proposed by small case series

ELIGIBILITY:
Inclusion Criteria:

* Patient gives an informed consent.
* Patient is over 18 years of age.
* Having a diagnosis of a primary dystonia confirmed by a trained movement disorders neurologist;
* Having failed or not tolerated conventional medical management, at the discretion of the neurologist managing the patient;

Exclusion Criteria:

* Having alternative diagnoses to a primary dystonic syndrome;
* Having comorbid neurodegenerative disorders that may affect mobility or cognition (e.g. comorbid Parkinson's disease);
* Having sequelae of prior brain insult (e.g. prior stroke or brain tumor);
* History of prior resectivebrain surgery (e.g. tumor resection);
* Not being a DBS candidate;
* Selection of alternative targets to conventional GPi;
* Receiving unilateral implants
* Having a higher surgical risk that precludes patient from having standard intraoperative mapping.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with dystonia, who have been cleared for DBS surgery or receiving a battery change who will receive the Percept battery.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Unified Dystonia Rating Scale (UDRS) | 12 months
  A clinical scale fo dystonia severity (0-4, 0:no symptoms, 4:extreme)
Burke-Fahn-Marsden Dystonia Rating Scale | 12 months
  A clinical scale fo dystonia severity (0-4, 0:no symptoms, 4:extreme)
Toronto Western Spasmodic Torticollis Rating Scale | 12 months
  A clinical scale of dystonia severity (0-4, 0:no symptoms, 4:extreme)

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gunduz, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States